CLINICAL TRIAL: NCT01639885
Title: Chemo-Immunotherapy, Gemcitabine With Pegylated Interferon Alpha-2b (Peg-Intron) With and Without p53 Synthetic Long Peptide (p53 SLP) Vaccine, for Patients With Platinum Resistant Ovarian Cancer CHIP Trial
Brief Title: Chemo-immunotherapy (Gemcitabine, Interferon-alpha 2b and p53 SLP) in Patients With Platinum-resistant Ovarian Cancer
Acronym: CHIP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, J.R. Kroep, MD phD, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHIP trial; 2010-023124-24 (EudraCT Number)
Record Dates: First submitted 2012-04-16; First posted 2012-07-13 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Recurrent Ovarian Cancer
Keywords: p53 overexpression; platinum-resistant
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Interferon alpha-2; p53 synthetic long peptide vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (No Intervention): Patients will receive standard care (gemcitabine)
- Group 2 (Experimental): Patients will receive standard care (gemcitabine) combined with interferon-alpha 2b (Peg-Intron)
  Interventions: Drug: Interferon Alfa-2b
- Group 3 (Experimental): Patients will receive standard care (gemcitabine) combined with interferon-alpha 2b (Peg-Intron) and p53 SLP vaccin
  Interventions: Drug: Interferon Alfa-2b; Biological: p53 SLP

INTERVENTIONS:
Drug: Interferon Alfa-2b — 1ug/kg (max 100ug) 7 days before and 22 days after first treatment with gemcitabine
  Arms: Group 2
Drug: Interferon Alfa-2b — 1ug/kg (max 100ug) 7 days before and 22 days after first treatment with gemcitabine
  Arms: Group 3
Biological: p53 SLP — 8.2.3 The p53 SLP vaccine consists of 9 synthetic 25-30 amino acids long overlapping peptides, spanning amino acids 70-235 of the wt-p53 protein (patent number WO2008147186). Peptides are prepared at the GMP facility of the Department of Clinical Pharmacy and Toxicology of the LUMC. At the day of immunization peptides (0.3 mg/peptide) were dissolved in dimethyl sulfoxide (DMSO, final concentration 20%) admixed with 20 mM phosphate buffer (pH7.5) and emulsified with an equal volume of Montanide ISA-51.The vaccine (2.7mL) is administered subcutaneously.
  Arms: Group 3

SUMMARY:
This study investigates the feasibility and immunogenicity of the triple combination of gemcitabine, Peg-Intron and p53 SLP vaccination in patients with platinum-resistant ovarian cancer.

DETAILED DESCRIPTION:
Recurrent ovarian cancer has a dismal prognosis and there is a pressing need to identify more efficient therapies. Ovarian cancer is highly immunogenic and good survival is tightly linked to the presence of tumor-infiltrating T cells and the absence of immunosuppressive immune cells. This anti-tumor immune response might be primed by chemotherapy.

Gemcitabine has immune-modulatory properties in addition to its direct cytotoxic effect in platinum resistant ovarian cancer. Additionally, Peg-Intron allows the full maturation of dendritic cells, thereby enhancing the anti-tumor response. Moreover, the tumor-associated self-antigen p53 is commonly over-expressed in ovarian cancer and can serve as a target for immunotherapy. Therefore, chemo-immunotherapy with gemcitabine and Peg-Intron plus/minus p53 SLP vaccination seems an attractive treatment for recurrent, p53+ ovarian cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histological proven epithelial ovarian cancer, peritoneal cavity or fallopian tube cancer (inclusive mucinous or clear cell tumors)
* Tumor over-expressing p53
* Progression of disease or relapse after previous therapy with platinum
* Measurable disease (RECIST 1.1) or elevated CA125 > 2 times the upper limit of normal within 3 months and confirmed
* Age ≥ 18 years
* WHO performance status 0-2
* Adequate bone marrow function: WBC ≥ 3.0 x 109/l, neutrophils ≥ 1.5 x 109/l, platelets ≥ 100 x 109/l
* Adequate liver function: bilirubin ≤ 1.5 x upper limit of normal (UNL) range, ALAT and/or ASAT ≤ 2.5 x UNL, Alkaline Phosphatase ≤5 x UNL
* Adequate renal function: the calculated creatinine clearance should be ≥ 50 mL/min
* Survival expectation > 3 months
* Patients must be accessible for treatment and follow-up
* Written informed consent according to the local Ethics Committee requirements

Exclusion Criteria:

* Previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix.
* Serious other diseases as recent myocardial infarction, clinical signs of cardiac failure or clinically significant arrhythmias
* Known hypersensitivity reaction to any of the components of the treatment
* Pregnancy or lactating
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-08; Primary Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Feasibility (change in grade III and IV toxicity) and change in immunogenicity of the triple combination of gemcitabine, Peg-Intron and p53 SLP vaccination | Before treatment, after 2 months and after 6 months after start therapy
  During the trial we will measure the incidence and severity of all side effects (according to CTC version 4.0). The change in immunogenecity will be measured according to the induction of p53-specific T cells upon treatment.

SECONDARY OUTCOMES:
Clinical outcome (response (RECIST 1.1) | Before treatment, after 2 months and after 6 months after start therapy
  Clinical outcome will be tested by analyzing CA125 in sera and tumor size at CT (by RECIST 1.1)and time from start treatment until death
The effect of this new treatment combination on the immune system | Before treatment, after two months and after 6 months after treatment
  Changes in plasma signature and tumor tissue will be measured
progression free survival | Before treatment, after 2 months and after 6 months after start therapy
overall survival | Before treatment, after 2 months and after 6 months after start therapy

CONTACTS AND LOCATIONS:
Overall Officials: Judith R Kroep, MD, PhD, Principal Investigator — Leiden University Medical Center
Locations (1):
- Leiden University Medical Center, Leiden, Netherlands